CLINICAL TRIAL: NCT04901325
Title: Baricitinib in the Treatment of Adults With Pyoderma Gangrenosum (PG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alex Ortega Loayza, Associate Professor of Dermatology, School of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baricitinib for PG Treatment
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pyoderma Gangrenosum; Skin Diseases; Wound Heal; Pyoderma; Skin Ulcer
Keywords: Baricitinib; JAK Kinase Inhibitors
MeSH Terms: conditions — Pyoderma Gangrenosum; Skin Diseases; Pyoderma; Skin Ulcer | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baricitinib for PG (Experimental): Subjects with PG will be treated with 4 mg once daily of baricitinib for 24 weeks in addition to starting stable dose (at least 2 weeks) of prednisone at 30 mg daily. Prednisone will be tapered based on a pre-established algorithm assessed by investigator.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Subjects with PG will be treated with 4 mg once daily of baricitinib for 24 weeks.
  Other Names: Olumiant

SUMMARY:
An Open-Label, Proof-Of-Concept, Study of Baricitinib for the Treatment of Pyoderma Gangrenosum

DETAILED DESCRIPTION:
This is a Phase II study that will be open label and include a total of 20 patients who will receive the investigational product. PG will be defined by the investigator and a second reviewer on the basis of results from clinical, histological and laboratory assessments. These patients will undergo 24 weeks of baricitinib dosed daily and stable dose of prednisone dosed daily with follow-up until week 36.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with study procedures/requirements
* Capable of giving informed consent
* Diagnosis of at least one PG ulcer by clinical, histological and laboratory assessments with a minimum wound size of 4 cm2.
* Male age 18-99 who agree to not father a child or donate sperm while on study and at least 1 week following last dose of the study drug. If subject is a sexually active male and could cause a pregnancy, subject must be sure that female partner(s) are using birth control that works well or not have sex.
* Female age 18-99; either of non-childbearing potential or of childbearing potential who test negative for pregnancy and agree to use at least two reliable methods of birth control or remain abstinent during the study and for at least 1 week following the last dose of baricitinib.
* Classic PG defined as deep ulceration with undermining violaceous borders.
* Are candidate for systemic therapy. All participants will be taking and clinically stable 30 mg (same ulcer size) of prednisone fort least two weeks at the start of the study. Patients must have discontinued immunosuppressive therapies (cyclosporine, azathioprine, mycophenolate mofetil, methotrexate, apremilast, dapsone) due to inadequate response or intolerance for at least 4 weeks prior to beginning the study drug.
* Undergoing at least once a week standard of care wound care at home or wound care facility.
* Willingness to travel to Oregon Health and Science University (OHSU) for all study visits, or living >30 miles from OHSU and willing/able to participate in remote videoconferencing visits with access to a computer with internet and webcam capabilities.

Exclusion Criteria:

* Have history of malignancy or lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for < 5years.
* Patients with cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinomas who have had active disease within 3 years of screening for this study. Active, untreated, acute or chronic infection (such as untreated tuberculosis), or immunocompromised to an extent that such that participation in the study would pose an unacceptable risk to the subject. (Treated infections such as latent tuberculosis after completion of the appropriate therapy are not excluded.Patients currently on treatment for active TB with drugs such as strong OAT-3 inhibitors will be excluded from study)
* Clinically serious infection or received intravenous antibiotics for an infection, within 4 weeks of randomization.
* Active viral infection that, based on the investigator's clinical assessment, makes the subject and unsuitable candidate for the study.
* Positive for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
* Symptomatic herpes zoster infection within 12 weeks of screening or recurrent or disseminated (even a single episode) herpes zoster.
* Symptomatic herpes simplex at the time of randomization or disseminated (even a single episode) herpes simplex
* History of disseminated opportunistic infections (e.g., listeriosis and histoplasmosis).
* Have a history of venous thromboembolism (VTE), or are considered at high risk for VTE as deemed by the investigator, or have 2 or more of the following risk factors for VTE:

  1. Aged >65 years.
  2. Body mass index (BMI) >35 kg/m2.
  3. Oral contraceptive use and current smoker.
* Creatinine Clearance <30 mL/min
* Wound care debridement of any PG ulcer within 2 weeks.
* Intralesional corticosteroids within 4 weeks of screening.
* Previous exposure to a Janus kinase (JAK) inhibitor (ruxolitinib, tofacitinib, upadacitinib, filgotinib). For biologic therapies, the specific washout periods used will at least 4 weeks for anakinra, etanercept, infliximab, adalimumab, alefacept, golimumab, secukinumab, ixekizumab, risankizumab, guselkumab, tildrakizumab, canakinumab, ustekinumab and at least 24 weeks for rituximab or efalizumab.
* Patients who are currently on immunosuppressive therapies or have not discontinued them for at least 4 weeks.
* Clinically significant (per investigator's judgement) drug or alcohol abuse within the last 6 months preceding the Baseline Visit.
* Have a live vaccine within 12 weeks prior to baseline or intend to have a live vaccine during the course of study.
* Had any major surgery within 8 weeks prior to baseline or will require major surgery during the study, which in the opinion of the investigator would pose an unacceptable risk to the subject.
* Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting. Uncontrolled hypertension - confirmed systolic blood pressure >160 mmHg or diastolic blood pressure >100 mm Hg.
* Gastrointestinal (GI) perforation (other than appendicitis or penetrating injury), diverticulitis or significantly increased for GI perforation (within past 6 months) per investigator judgement; any condition could interfere with drug absorption including but not limited to short bowel syndrome.
* Presence of significant uncontrolled respiratory, hepatic, renal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of the data.
* Have clinical laboratory test results at screening that are outside the normal reference range of the population and are considered clinically significant, or have any of the following specific abnormalities: Neutrophil count <1500 cells/µL, lymphocyte count <500 cells/µL, platelet count <100,000 cells/µL, aspartate transaminase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal, hemoglobin <10 g/dL for male and female subjects, eGFR>60.
* Women who are lactating or breastfeeding.
* Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the investigator.
* Are investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling).
* Are currently enrolled in, or discontinued from a clinical trial involving an investigational product or non-approved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* History of myocardial infarction, stroke and New York Heart Association Stage II/IV heart failure
* Patients on concomitant medication with a Strong OAT-3 inhibitor for an existing condition will be excluded from study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Healing | Week 24
  defined as the proportion of patients with complete re-epithelization, defined as 100% re-epithelialization without any drainage, of the target ulcer at week 24.

SECONDARY OUTCOMES:
Physician Global Assessment (PGA) | Week 24
  Assessing the proportion of patients that show target ulcer healing in response to study treatment as measured by achieving PGA between 0 and 1 after treatment with baricitinib at week-36 52. This scale has been used in previous trials:
  1. 0 = total resolution of target ulcer with no signs of active PG
  2. 1= almost completely healed target ulcer with only minimal signs of active PG
  3. 2 = evidence of target ulcer healing which involves at least 50% of ulcer/ulcer margin
  4. 3 = evidence of target ulcer healing which involves less than 50% of ulcer/margin
  5. 4 = no evidence of target healing ulcer
Percent change in lesion surface area | Week 0 and 24
  The percent change in surface area of target lesion of PG (two-dimensional surface in cm²) using digital photography and acetate tracing at Week 0 and Week 24
Mean change in lesion surface area | Week 0 and 24
  The mean change in surface area of target lesion of PG (two-dimensional surface in cm²) using digital photography and acetate tracing
Mean change in Physician Global Assessment (PGA) | Week 0 and 24
  The mean change in Physician global assessment (PGA) 5-point scale at week 0 to week 24
Sustained healing | Week 36
  The proportion of patients with target ulcer that remains healed by week 36
Decrease in ulcer area size | Week 24
  The proportion of patients with decrease in ulcer area size of at least 50% after treatment at week 24
Time to healing | Over 36-week period of study.
  Time to which sterile dressings are not required.
Time to recurrence (weeks) | 36 weeks
  Interval between target lesion healing and further episodes of PG at any site through the study.
Number of treatment failures | By week 24
  Treatment intolerance, number of patients switching into standard of care or target lesion unhealed.
Adverse reactions to medications | Over 24-week period of study.
  Possibly-, probably- or related throughout the study.
Quality of life change (as measured by the Dermatology Life Quality Index) | Week 24
  Proportion of subjects achieving a 4-point change in quality of life measured by the Dermatology Life Quality Index (DLQI) at week 24, and mean change in DLQI score at week 24. The DLQI is a validated tool for inflammatory skin conditions. It is a 10-question survey, scored 0 - 30 points. For inflammatory skin conditions, a 4-point change in DLQI score is considered clinically important.
Mean change in quality of life (measured by Dermatology Life Quality Index) | Week 0 and 24
  Mean change in DLQI score from week 0 to week-24.
Skin pain scale | Week 0 to 24
  The proportion of patients with a 2 point decrease in the point numeric pain rating scale (NRS) at week 0 and week-24. The pain NRS is a subject-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable."

OTHER OUTCOMES:
Evaluation of cytokine gene expression | Week 0 and week 24
  15. Evaluation of cytokine gene expression before and after treatment in skin, wound fluid, saliva and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Alex G Ortega-Loayza, MD, MCR, Principal Investigator — Oregon Health & Science University, Department of Dermatology
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braswell SF, Kostopoulos TC, Ortega-Loayza AG. Pathophysiology of pyoderma gangrenosum (PG): an updated review. J Am Acad Dermatol. 2015 Oct;73(4):691-8. doi: 10.1016/j.jaad.2015.06.021. Epub 2015 Aug 5. PMID 26253362
- [Background] Alves de Medeiros AK, Speeckaert R, Desmet E, Van Gele M, De Schepper S, Lambert J. JAK3 as an Emerging Target for Topical Treatment of Inflammatory Skin Diseases. PLoS One. 2016 Oct 6;11(10):e0164080. doi: 10.1371/journal.pone.0164080. eCollection 2016. PMID 27711196
- [Background] Shanmugam VK, McNish S, Shara N, Hubley KJ, Kallakury B, Dunning DM, Attinger CE, Steinberg JS. Chronic leg ulceration associated with polycythemia vera responding to ruxolitinib (Jakafi((R))). J Foot Ankle Surg. 2013 Nov-Dec;52(6):781-5. doi: 10.1053/j.jfas.2013.07.003. Epub 2013 Aug 14. PMID 23953278
- [Background] Nasifoglu S, Heinrich B, Welzel J. Successful therapy for pyoderma gangrenosum with a Janus kinase 2 inhibitor. Br J Dermatol. 2018 Aug;179(2):504-505. doi: 10.1111/bjd.16468. Epub 2018 May 21. No abstract available. PMID 29451690
- [Background] Kochar B, Herfarth N, Mamie C, Navarini AA, Scharl M, Herfarth HH. Tofacitinib for the Treatment of Pyoderma Gangrenosum. Clin Gastroenterol Hepatol. 2019 Apr;17(5):991-993. doi: 10.1016/j.cgh.2018.10.047. Epub 2018 Nov 4. PMID 30404036
- [Background] Palanivel JA, Macbeth AE, Levell NJ. Pyoderma gangrenosum in association with Janus kinase 2 (JAK2V617F) mutation. Clin Exp Dermatol. 2013 Jan;38(1):44-6. doi: 10.1111/j.1365-2230.2012.04375.x. Epub 2012 May 21. PMID 22607468
- [Background] Ortega-Loayza AG, Nugent WH, Lucero OM, Washington SL, Nunley JR, Walsh SW. Dysregulation of inflammatory gene expression in lesional and nonlesional skin of patients with pyoderma gangrenosum. Br J Dermatol. 2018 Jan;178(1):e35-e36. doi: 10.1111/bjd.15837. Epub 2017 Dec 5. No abstract available. PMID 28734003
- [Background] Liu D, Ahmet A, Ward L, Krishnamoorthy P, Mandelcorn ED, Leigh R, Brown JP, Cohen A, Kim H. A practical guide to the monitoring and management of the complications of systemic corticosteroid therapy. Allergy Asthma Clin Immunol. 2013 Aug 15;9(1):30. doi: 10.1186/1710-1492-9-30. PMID 23947590
- [Background] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772